CLINICAL TRIAL: NCT01311518
Title: A Randomized, Double-blind, Placebo-Controlled, Study of the Safety and Efficacy of RGN-352 in Subjects With an Acute ST Elevation Myocardial Infarction (STEMI) After Occlusion of the Proximal Left Anterior Descending Coronary Artery
Brief Title: A Study of the Safety and Efficacy of Injectable Thymosin Beta 4 for Treating Acute Myocardial Infarction
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial never initiated
Sponsor: RegeneRx Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-MI-201
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Acute Myocardial Infarction; ST Elevation Myocardial Infarction; STEMI
Keywords: Thymosin Beta 4; Thymosin β4 (Tβ4) Injectable Solution; RGN-352
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — thymosin beta(4)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Drug: Placebo
- Drug: Thymosin Beta 4 injectable (Active Comparator)
  Interventions: Drug: Drug: Injectable Thymosin beta 4

INTERVENTIONS:
Drug: Drug: Placebo — Injectable administration by slow intravenous bolus, 0.00% Thymosin Beta 4 daily for 3 days then weekly for 4 consecutive weeks
  Other Names: 0.00% Thymosin Beta 4
  Arms: Placebo
Drug: Drug: Injectable Thymosin beta 4 — Injectable administration of Thymosin Beta 4 by intravenous bolus at 1200 mg, or 450 mg daily for 3 days then weekly for 4 consecutive weeks
  Other Names: Injectable Thymosin Beta 4; Tβ4 Injectable Solution; RGN-352
  Arms: Drug: Thymosin Beta 4 injectable

SUMMARY:
The objective of this study is to evaluate the safety and tolerability of two active doses of RGN-352 (thymosin beta 4, Tβ4, Injectable Solution) in patients with acute myocardial infarction receiving percutaneous coronary intervention angioplasty with or without stent placement. Approximately 75 subjects will be randomized to receive one of two RGN-352 doses of 1200 mg, or 450 mg, or placebo, administered iv by iv push daily for the first 3 consecutive days and weekly for 4 more weeks.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled, parallel-group, dose finding study. Eligible subjects will be randomized to receive one of two doses of RGN-352 or matching placebo with an equal allocation ratio (i.e., 1:1:1). Approximately 75 subjects will be randomized to study treatment to achieve at least 60 evaluable subjects with 20 to 25 subjects per group. Subjects will be randomized to receive one of two RGN-352 doses of 1200 mg, or 450 mg, or placebo, administered iv by iv push daily for the first 3 consecutive days and weekly for 4 consecutive weeks. Study subjects will undergo cardiac angiography to assess initial coronary artery patency and Thrombolysis In Myocardial Infarction flow grade both pre- and post-percutaneous coronary intervention (PCI) angioplasty. A total of 7 doses will be administrated over the treatment period. The first dose of either RGN-352 or placebo will be administered to randomized subjects following PCI angioplasty and specifically within 30 minutes after balloon deflation, with a further 2 doses. The remaining 4 doses will be given weekly for 4 consecutive weeks. Follow-up is on Months 2, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects
2. Negative urine pregnancy test at Screening
3. An electrocardiogram
4. First acute anterior MI
5. Baseline angiography
6. Onset of chest pain symptoms to initial PCI angioplasty time is 2 to 6 hours
7. Written informed consent reviewed and signed by the subject or legally authorized representatives

Exclusion Criteria:

1. Intention to treat subject with thrombolytic therapy following assertion of Thrombolysis In Myocardial Infarction(TIMI) flow 0 or 1 during qualifying angiogram
2. History of Myocardial infarctionI or congestive heart failure
3. Non-atherosclerotic etiology of acute myocardial infarction
4. Cardiogenic shock (systolic blood pressure <90 despite adequate left ventricle filling pressure or requiring catecholamines) or other hemodynamic instability at baseline
5. Further transcatheter or surgical revascularization, e.g., coronary artery bypass graft planned per baseline angiogram
6. Lactating women
7. Past or present evidence of malignancy
8. Women who have had menarche but have not completed menopause, have not been surgically sterilized (bilateral tubal ligation or hysterectomy), do not have a partner with documented sterility (including vasectomy), or are not using adequate contraception (combined hormonal or double-barrier method of contraception, or sexual abstinence are the only methods of contraception acceptable for this study)
9. Ongoing infectious disease including human immunodeficiency virus (HIV) and hepatitis
10. Clinically significant respiratory, renal, metabolic, liver, central nervous system or other comorbid disease, except current cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Total MRI infarct zone derived from cardiac MRI scan | Day 28

SECONDARY OUTCOMES:
MRI-derived myocardial salvage index, mass, Left Ventricle (LV) ejection fraction,systolic and end diastolic volumes | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: J.J. Finkelstein, BBA, Study Director — RegeneRx Biopharmaceuticals, Inc.